CLINICAL TRIAL: NCT00990561
Title: A Clinical Study Comparing the Efficacy of Ultravate Ointment Once Daily vs. Twice Daily in Combination With Lac-Hydrin Lotion in the Treatment of Stable Plaque Psoriasis
Brief Title: Comparing the Efficacy of Ultravate Ointment in Combination With Lac-Hydrin Lotion in the Treatment of Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ultravate Lac-Hydrin Ranbaxy; H5939-34434-01
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Stable Plaque Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Twice Daily Ultravate (Active Comparator): Patients will apply both Ultravate ointment and LacHydrin lotion twice daily
  Interventions: Drug: Ultravate ointment twice daily + LacHydrin lotion twice daily
- Once daily Ultravate (Active Comparator): Patients will apply Ultravate ointment once daily, but will use LacHydrin lotion twice daily
  Interventions: Drug: Ultravate ointment once daily + LacHydrin lotion twice daily

INTERVENTIONS:
Drug: Ultravate ointment twice daily + LacHydrin lotion twice daily — Topical corticosteroid
  Other Names: Halobetasol ointment, Ammonium lactate lotion
  Arms: Twice Daily Ultravate
Drug: Ultravate ointment once daily + LacHydrin lotion twice daily — Topical corticosteroid
  Other Names: Halobetasol ointment, Ammonium lactate lotion
  Arms: Once daily Ultravate

SUMMARY:
This is an investigator-masked, randomized, parallel, clinical study comparing the efficacy of once daily versus twice daily application of Ultravate® ointment (halobetasol propionate 0.05% ointment) in combination with Lac-Hydrin lotion (ammonium lactate topical) in the treatment of stable plaque psoriasis. 1) Phase 1: Patients will be treated for two weeks with combination therapy using Ultravate® ointment with Lac-Hydrin lotion and their psoriasis plaques will be evaluated to test efficacy of the medication. Half the subjects will be randomized to receive treatment with once a day Ultravate® ointment and twice daily Lac-Hydrin lotion; the other half of subjects will receive twice daily Ultravate® ointment with twice daily Lac-Hydrin lotion. Ultravate® ointment will be discontinued following two weeks of treatment, in compliance with its FDA indication. Phase 2: The second treatment phase will consist of a four-week observation period. Subjects will be re-randomized to either continue using twice daily Lac-Hydrin lotion, versus no treatment. The purpose of this second phase of the study is to investigate whether use of Lac-Hydrin monotherapy twice daily can minimize risk of recurrence and maximize duration of therapeutic effect. Part of this clinical study consists of the use of patient and physician satisfaction questionnaires. These questionnaires will include questions about the satisfaction with the formulation of each agent, questions about compliance with treatment, etc. Such questions could be used to demonstrate patient and physician satisfaction with each agent, with combination therapy, and to compare patient satisfaction rates among those randomized to once daily versus twice daily application of Ultravate® ointment. The hypothesis is that Ultravate ointment once daily in combination with Lac-Hydrin twice daily is equal in efficacy to Ultravate ointment twice daily in combination with Lac-Hydrin twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed by an investigator to have stable plaque psoriasis with no more than 10% body surface area involvement.
* A subject must have an overall baseline score of 6 (moderate) or greater based on a twelve-point scale on the Psoriasis Severity Assessment (PSA) form. Elevation, erythema, and scale will each be graded on a four point scale with a maximum total of 12 points. Each of these 3 variables should be scored as at least a two. (Plaque elevation is defined as the total elevation, including adherent scales, relative to the surrounding skin).
* For female patients of childbearing potential, a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation).
* Negative urine pregnancy test at the time of study entry (for female patients of childbearing potential).
* Written, informed consent and photographic release.
* Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* A female subject who is pregnant, nursing an infant or planning a pregnancy during the study (throughout the course of the study, women of childbearing potential must use reliable forms of contraception [i.e., abstinence, spermicides, condoms, or other reliable forms of contraception other than oral contraceptives].
* A subject with any uncontrolled systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
* A subject with the presence of any skin disease that might interfere with the diagnosis or evaluation of the test medications.
* A subject that has a condition or is in a situation which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.
* A subject with spontaneously improving or rapidly deteriorating plaque psoriasis.
* A subject with pustular or erythrodermic psoriasis.
* A subject diagnosed by an investigator to have stable plaque psoriasis involvement that exceeds more than 10% of the subject's body surface area.
* Use of systemic agents such as oral retinoids, methotrexate, cyclosporine or systemic corticosteroids within four weeks prior to study entry.
* Use of biologic agents such as alefacept, infliximab, efalizumab, adalimumab, or etanercept within four weeks prior to study entry.
* Use of topical drugs that might alter the course of psoriasis (e.g., corticosteroids, retinoids, vitamin D analogues, salicylic acid, tacrolimus, tar and anthralin,) or has received Ultraviolet B treatment within two weeks prior to study entry.
* Use of phototherapy with psoralen ultraviolet A treatment within four weeks prior to study entry.
* A subject with a known sensitivity to any of the study treatments and/or their components.
* A subject who will require excessive or prolonged exposure to ultraviolet light (e.g., sunlight, tanning beds) during the study.
* A subject who anticipates a need to use other topical or systemic therapy that might alter the course of psoriasis.
* A subject who anticipates the need for surgery or hospitalization during the study.
* Concurrent involvement in any other clinical study with an investigational drug or device, or participation in a clinical study within 30 days prior to entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Bhutani, MD, Study Director — UCSF Clinical Fellow
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from our medical clinic as well as through flyers posted at other University of California at San Francisco sites.
Pre-assignment Details: Patients were required to have a 2 week washout from topicals, 1 month washout from any systemic agents.
Period: Period 1
Arm/Group | Twice Daily Topical Ultravate Ointment + LacHyrin Twice Daily | Once Daily Topical Ultravate Ointment + LacHydrin Lotion | Lac-Hydrin Topically Twice a Day | No Treatment
Started | 20 | 20 | 0 | 0
Completed | 20 | 19 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Twice Daily Topical Ultravate Ointment + LacHyrin Twice Daily | Once Daily Topical Ultravate Ointment + LacHydrin Lotion | Lac-Hydrin Topically Twice a Day | No Treatment
Started | 0 | 0 | 20 | 19
Completed | 0 | 0 | 20 | 17
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ultravate Once a Day: Ultravate ointment applied once daily
- Total: Total of all reporting groups
Arm/Group | Ultravate Twice a Day | Ultravate Once a Day | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: Years] | NA [NA to NA] — Age was not analyzed by sub-group. Just overall. | NA [NA to NA] — Age was not analyzed by sub-group. Just overall. | 44.2 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Psoriasis Area Severity Index (PASI) Score
Description: PASI is a scale that measures psoriasis severity based on erythema, induration, scaling, and body surface area covered. It ranges from 0 (no disease) to 72 (most extensive).
Time Frame: 2 weeks
Population: This was a pilot study and the number was based on the available budget to perform the study.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Ultravate 0.05% Ointment Twice Daily: Ultravate twice daily to affected area.
- Ultravate 0.05% Ointment Once Daily: Ultravate one daily to affected area.
Arm/Group | Ultravate 0.05% Ointment Twice Daily | Ultravate 0.05% Ointment Once Daily
Number analyzed (Participants) | 20 | 20
units on a scale | 2.6 [2.6 to 3.1] | 3 [2.4 to 3.5]
Statistical Analysis 1: Comparison: Ultravate 0.05% Ointment Twice Daily; Null hypothesis = there is no difference between using ultravate once daily vs. twice daily; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 3.0

ADVERSE EVENTS:
Arm/Group | Ultravate Twice a Day | Ultravate Once a Day
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No